CLINICAL TRIAL: NCT06912867
Title: The BRAVE-CAN Study: A Clinical Trial Investigating the Effects of Blood Flow Restriction Training on Lower Extremity Muscle Strength, Muscle Thickness, and Sport Motivation in Adolescent Male National Canoe Athletes
Brief Title: Effects of BFR Training on Muscle Strength, Thickness, and Motivation in National Adolescent Male Canoe Athletes
Acronym: BRAVE-CAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Burçin Uğur Tosun, Principal Investigator PhD Physiotherapist Burcin Ugur Tosun, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2025-43
Record Dates: First submitted 2025-03-27; First posted 2025-04-06 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Muscle Strength; Muscle Hypertrophy; Sport Performance
Keywords: Blood Flow Restriction; Muscle Strength; Adolescent Athletes; Canoe Sprint; Sport Motivation

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned into two groups using block randomization: an intervention group receiving blood flow restriction (BFR) training and a control group continuing regular training without BFR. Both groups followed their respective training protocols over an 8-week period. Outcomes were assessed pre- and post-intervention by blinded evaluators.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors were blinded to group allocation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BFR Training Group (Experimental): Participants performed supervised low-load resistance training with BFR using KAATSU C3 equipment twice a week for 8 weeks.
  Interventions: Behavioral: Blood Flow Restriction (BFR) Exercise Program
- Control Group (No Intervention): Participants in this group continued their standard canoe training program without additional blood flow restriction exercises.

INTERVENTIONS:
Behavioral: Blood Flow Restriction (BFR) Exercise Program — Participants performed supervised low-load resistance training with BFR using KAATSU C3 equipment twice a week for 8 weeks.
  Arms: BFR Training Group

SUMMARY:
The aim of this study is to evaluate the effects of blood flow restriction (BFR) exercises on lower extremity muscle strength, muscle thickness, and sport-specific motivation in adolescent elite male canoe athletes. Participants aged 15-18 years will perform low-intensity resistance exercises supported by BFR twice a week for 8 weeks. Pre- and post-intervention measurements will include one-repetition maximum (1RM) for muscle strength, ultrasound for muscle thickness, and the Sport Motivation Scale for assessing motivation. Findings are expected to contribute to optimizing training protocols for canoe athletes and to reveal the potential performance-enhancing role of BFR training.

DETAILED DESCRIPTION:
This randomized controlled trial aims to investigate the physiological and psychological effects of blood flow restriction (BFR) training on adolescent elite male canoe athletes. Canoeing is a demanding endurance sport requiring well-developed upper and lower extremity strength, core stability, and high levels of sport-specific motivation. In adolescent athletes, whose musculoskeletal and hormonal systems are still developing, traditional high-load resistance training may not always be feasible or safe. BFR training, which involves restricting venous blood flow while performing low-intensity exercises, has emerged as a potential alternative for promoting muscle hypertrophy and strength with reduced mechanical stress.

In this study, a total of 40 adolescent male canoe athletes aged 15 to 18 years are enrolled and randomized into two groups: a BFR intervention group (n=28) and a control group (n=12). The intervention group participates in a supervised BFR-supported resistance training program twice a week for 8 weeks using KAATSU C3 equipment applied to the lower limbs. Both groups continue their regular canoe training programs. Assessments are performed before and after the 8-week training period by blinded evaluators.

Primary outcome measures include isokinetic muscle strength tests, ultrasound-based measurements of muscle thickness and cross-sectional area (CSA), and scores from the validated Sport Motivation Scale. The study is designed to explore potential effects of BFR training on muscular strength, hypertrophy, sprint capacity, and motivational subdomains in this athletic population.

This research aims to contribute to the growing body of literature regarding the applicability of BFR training in adolescent athletes, with a focus on its physiological and psychological outcomes. Findings from this study may help inform future training strategies for youth involved in high-performance sports.

ELIGIBILITY:
Inclusion Criteria:

* Male athletes aged between 15 and 18 years
* Registered elite-level canoe athletes actively training within a national program
* Minimum of 2 years of canoe sport experience
* Voluntary participation with informed consent (for minors: parental/guardian consent)
* Medically cleared to participate in physical training and testing

Exclusion Criteria:

* Existing orthopedic injuries or musculoskeletal disorders affecting lower extremities
* History of cardiovascular, neurological, or metabolic diseases
* Non-compliance with the training protocol during the study
* Participation in any other structured strength training program during the study period
* Use of medications or supplements affecting muscle performance or motivation

Ages: 15 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-10 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Lower Extremity Muscle Strength (Peak Torque, Nm) - measured via isokinetic dynamometry | Baseline (Week 0) and Post-intervention (Week 8)
  Muscle strength of the quadriceps and hamstring muscles was assessed using an isokinetic dynamometer (Biodex System 4) at angular velocities of 60°/s and 300°/s. Peak torque (in Newton-meters) was recorded for both right and left lower limbs. Measurements were conducted at baseline and after the 8-week intervention period by a blinded physiotherapist.
Muscle Thickness (mm) - measured via ultrasound | Baseline (Week 0) and Post-intervention (Week 8)
  Muscle thickness and cross-sectional area of the quadriceps femoris and hamstring muscle groups were evaluated using B-mode ultrasound imaging (Mindray DP-10). Measurements were taken bilaterally from standardized anatomical landmarks in a resting position. The assessment was performed by a blinded sports medicine physician at baseline and after 8 weeks of training.
Sport-Specific Motivation Score - measured using the Sport Motivation Scale (validated Turkish version) | Baseline (Week 0) and Post-intervention (Week 8)
  Sport-specific motivation levels will be assessed using the Turkish-validated version of the Sport Motivation Scale-II. The scale consists of 18 items rated on a 7-point Likert scale ranging from 1 (Does not correspond at all) to 7 (Corresponds exactly). Total scores range from 18 to 126, with higher scores indicating greater overall sport motivation.
  The scale includes three subdimensions relevant to this study:
  Motivation to Show Strength
  Motivation to Approach Success
  Motivation to Avoid Failure Subscale scores are calculated as the mean of related items. Higher subscale scores indicate a stronger level of that specific motivational trait.

CONTACTS AND LOCATIONS:
Overall Officials: burcin ugur tosun, PHD, Principal Investigator — "Bandırma Onyedi Eylül University, Faculty of Health Sciences"
Locations (1):
- Burcin Ugur Tosun, Famagusta, Cyprus